CLINICAL TRIAL: NCT01314443
Title: Cardioprotective Synergy of Smoking Cessation and γ-Tocopherol in Restoring Vascular Endothelial Function
Brief Title: Impact of Smoking Cessation and γ-Tocopherol to Restore Vascular Endothelial Function
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Connecticut (Other)
Responsible Party: Principal Investigator, Richard Bruno, Associate Professor, University of Connecticut
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Basic Science
Other Study IDs: H10-212
Record Dates: First submitted 2011-03-10; First posted 2011-03-14 (Estimated); Results first posted 2013-03-06 (Estimated); Last update posted 2015-01-21 (Estimated); Status verified 2015-01

CONDITIONS: Endothelial Dysfunction
Keywords: smoking cessation; gamma-tocopherol; nicotine-replacement therapy; oxidative stress
MeSH Terms: conditions — Smoking Cessation | interventions — Nicotine Replacement Therapy; Tobacco Use Cessation Devices; Nicotine; gamma-Tocopherol; Vitamin E; Corn Oil

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo + Smoking Cessation (Experimental): Individuals will quit smoking without use of nicotine replacement therapy (NRT) and ingest a placebo for 7 days
  Interventions: Other: Placebo; Behavioral: Smoking cessation
- Supplement + Smoking Cessation (Experimental): Individuals will quit smoking without the use of nicotine replacement therapy (NRT) and ingest a gamma-tocopherol supplement for 7 days
  Interventions: Dietary Supplement: Gamma-Tocopherol; Behavioral: Smoking cessation
- Placebo + Nicotine Replacement Therapy (Experimental): Individuals will quit smoking with the use of nicotine replacement therapy (NRT) and ingest a placebo for 7 days
  Interventions: Other: Nicotine Replacement Therapy (NRT); Other: Placebo
- Supplement+Nicotine Replacement Therapy (Experimental): Individuals will quit smoking with the use of nicotine replacement therapy (NRT) and ingest a gamma-tocopherol supplement for 7 days
  Interventions: Other: Nicotine Replacement Therapy (NRT); Dietary Supplement: Gamma-Tocopherol

INTERVENTIONS:
Other: Nicotine Replacement Therapy (NRT) — Participants will quit smoking with nicotine patches
  Other Names: Nicotine patches; NicoDerm
  Arms: Placebo + Nicotine Replacement Therapy; Supplement+Nicotine Replacement Therapy
Dietary Supplement: Gamma-Tocopherol — Participants will take gamma-tocopherol (500 mg/d) supplements for 7 days
  Other Names: Vitamin E
  Arms: Supplement + Smoking Cessation; Supplement+Nicotine Replacement Therapy
Other: Placebo — Participants will take placebo for 7 days
  Other Names: Corn oil
  Arms: Placebo + Nicotine Replacement Therapy; Placebo + Smoking Cessation
Behavioral: Smoking cessation — Participants will quit smoking without any pharmacological aids
  Arms: Placebo + Smoking Cessation; Supplement + Smoking Cessation

SUMMARY:
Cigarette smoking is a significant risk factor for cardiovascular disease (CVD) and is the leading cause of premature mortality in the US. The detrimental effects of smoking on vascular dysfunction are attributed to the effects of smoke itself and the inflammatory responses it induces. Smoking cessation restores vascular function by alleviating these stress responses. However, smoking cessation with nicotine replacement therapy (NRT), the prevailing approach to mitigate tobacco dependence, fails to allow full restoration of vascular function. Thus, a critical public health problem exists to understand how NRT prevents restoration of vascular function and how these NRT-mediated impairments can be overcome by using gamma-tocopherol (g-T) as an innovative co-therapy. The objective of this study is to conduct a clinical intervention trial that aims to reduce CVD risk by defining how smoking cessation and g-T restore vascular function. The hypothesis is that smoking cessation and dietary g-T supplementation will synergistically restore smoking-induced impairments in vascular function by ameliorating oxidative/nitrosative stress responses, and that g-T will facilitate full restoration of vascular function otherwise precluded by NRT. A placebo-controlled, g-T intervention study will be conducted in cigarette smokers undergoing nicotine-free or NRT smoking cessation. Prior to and after 24 h and 7 days of placebo or g-T administration, vascular function will be evaluated using a non-invasive ultrasound technique and an array of antioxidants and biomarkers for vascular inflammation and oxidative/nitrosative stress responses will be assessed. Collectively, these studies will help identify how vascular function is regulated in individuals undergoing smoking cessation, and whether g-T can be used as a strategy to better improve vascular function during smoking cessation.

DETAILED DESCRIPTION:
While it is well known that smoking cessation reduces the risk of cardiovascular disease (CVD), the rate in which CVD risk is normalized is relatively slow. This suggests a need to better define co-therapies that target oxidative stress and inflammatory responses that otherwise impair vascular function. In this randomized placebo-controlled clinical study, smokers undergoing smoking cessation with or without nicotine replacement therapy will receive dietary supplementation of gamma-tocopherol (500 mg/day) or placebo for 7 days. Their vascular function and biomarkers of CVD risk (inflammatory proteins, antioxidants, oxidized lipids) will be assessed prior to, and at 1 day and 7 days during smoking cessation with and without gamma-tocopherol supplementation to define potential mechanisms by which gamma-tocopherol may accelerate the restoration of vascular function and assist in reducing CVD risk.

ELIGIBILITY:
Inclusion Criteria:

* male or female between 18-60 y,
* premenopausal status for women
* healthy, verified by serum clinical chemistry
* stable body weight (±5 lbs) for 2-mo and BMI 19-30 kg/m2
* non-nutritional supplement user for >2-mo
* free of known diseases including diabetes, CVD, cancer, infections, HIV/AIDS, hepatitis, and bleeding disorders
* resting blood pressure <140/90 mm Hg;
* smokers (≥10 cigarettes/d, ≥1 year)
* maintaining normal exercise patterns (<7 h/week) and willingness to avoid exercise 24 h prior to blood sampling and vascular testing
* willingness to ingest a dietary vitamin E supplement (gamma-tocopherol; 500 mg/d) or a placebo (composed of tocopherol-free corn oil) daily for 1 week.

Exclusion Criteria:

* serum chemistry outside normal limits
* alcohol consumption >3 drinks/d or >10 drinks per week
* nutritional supplement user with past 2 months
* >7 hours/week of exercise
* use of any pharmacological therapy to treat high cholesterol or high blood pressure
* pregnancy, lactation, or initiation or change in hormonal birth control within the previous 3 mo
* use of vasoactive compounds (e.g. erectile dysfunction medication, omega 3-fatty acids, niacin)
* suffering from major psychiatric illnesses
* currently using non-nicotine aids or drugs to quit smoking; or 10) allergy to adhesive tape.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 67 (Actual)
Dates: Start 2011-01; Primary Completion 2011-11 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard S Bruno, PhD, RD, Principal Investigator — University of Connecticut
Locations (1):
- University of Connecticut, Storrs, Connecticut, United States

REFERENCES:
- [Result] Mah E, Pei R, Guo Y, Ballard KD, Barker T, Rogers VE, Parker BA, Taylor AW, Traber MG, Volek JS, Bruno RS. gamma-Tocopherol-rich supplementation additively improves vascular endothelial function during smoking cessation. Free Radic Biol Med. 2013 Dec;65:1291-1299. doi: 10.1016/j.freeradbiomed.2013.09.016. Epub 2013 Sep 27. PMID 24075893
- [Derived] Mah E, Pei R, Guo Y, Masterjohn C, Ballard KD, Taylor BA, Taylor AW, Traber MG, Volek JS, Bruno RS. Greater gamma-tocopherol status during acute smoking abstinence with nicotine replacement therapy improved vascular endothelial function by decreasing 8-iso-15(S)-prostaglandin F2alpha. Exp Biol Med (Maywood). 2015 Apr;240(4):527-33. doi: 10.1177/1535370214556948. Epub 2014 Oct 30. PMID 25361769

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment took place in and around the community surrounding the University of Connecticut. Recruitment occurred from 2010-2011.
Pre-assignment Details: Health status of participants was determined from a comprehensive metabolic panel as well as circulating lipid levels. Individuals having serum chemistries outside of acceptable limits were not enrolled.
Groups:
- Dietary Supplement + Smoking Cessation: Individuals will ingest gamma-tocopherol (500 mg/d) for 7 days while undergoing smoking cessation without any aids
- Placebo + Smoking Cessation: Individuals will ingest placebo for 7 days while undergoing smoking cessation without any aids
- Dietary Supplement + Nicotine Replacement Therapy: Individuals will ingest gamma-tocopherol (500 mg/d) for 7 days while undergoing smoking cessation with the use of nicotine replacement therapy
- Placebo + Nicotine Replacement Therapy: Individuals will ingest placebo for 7 days while undergoing smoking cessation with the use of nicotine replacement therapy
Period: Overall Study
Arm/Group | Dietary Supplement + Smoking Cessation | Placebo + Smoking Cessation | Dietary Supplement + Nicotine Replacement Therapy | Placebo + Nicotine Replacement Therapy
Started | 18 | 19 | 15 | 15
Completed | 14 | 16 | 13 | 13
Not Completed | 4 | 3 | 2 | 2
Not completed — Withdrawal by Subject | 2 | 1 | 1 | 1
Not completed — Protocol Violation | 2 | 2 | 1 | 1

BASELINE CHARACTERISTICS:
Population: 11 participants from the 67 participants enrolled in the study were excluded from all analysis (including baseline). Five participants withdrew from the study before completion and six participants were identified as non-compliant and were removed from the study. Thus, baseline analysis was performed on the remaining 56 participants.
Groups:
- Supplement + Smoking Cessation: Individuals will ingest gamma-tocopherol (500 mg/d) for 7 days while undergoing smoking cessation without any aids
- Supplement + Nicotine Replacement Therapy: Individuals will ingest gamma-tocopherol (500 mg/d) for 7 days while undergoing smoking cessation with the use of NRT
- Placebo + Nicotine Replacement Therapy: Individuals will ingest placebo for 7 days while undergoing smoking cessation with the use of NRT
- Total: Total of all reporting groups
Arm/Group | Supplement + Smoking Cessation | Placebo + Smoking Cessation | Supplement + Nicotine Replacement Therapy | Placebo + Nicotine Replacement Therapy | Total
Number analyzed (Participants) | 14 | 16 | 13 | 13 | 56
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 14 | 16 | 13 | 13 | 56
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 22 (4) | 22 (4) | 26 (8) | 25 (8) | 24 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 5 | 4 | 19
  Male | 9 | 11 | 8 | 9 | 37
Region of Enrollment [Number; unit: participants]
  United States | 14 | 16 | 13 | 13 | 56

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change in Brachial Artery Flow-mediated Dilation at Day 7 From Day 0
Description: Flow-mediated dilation (FMD) of the brachial artery is measured to assess vascular endothelial function. FMD is obtained by monitoring change in vessel diameter before and after brachial artery occlusion with a blood pressure cuff. The unit of FMD is % and is calculated using the following equation: FMD = [(peak dilation at post occlusion - vessel diameter at preocclusion)/vessel diameter at preocclusion]*100.
Time Frame: Day 0 and 7 of intervention
Population: Analysis was performed on all participants completing the 7 d intervention
Measure: Mean (Standard Error); unit: % of preocclusion diameter
Arm/Group | Dietary Supplement + Smoking Cessation | Placebo + Smoking Cessation | Dietary Supplement + Nicotine Replacement Therapy | Placebo + Nicotine Replacement Therapy
Number analyzed (Participants) | 14 | 16 | 13 | 13
% of preocclusion diameter | 4.08 (0.61) | 2.77 (0.35) | 2.97 (0.51) | 2.66 (0.44)

2. Secondary Outcome: Absolute Change From Baseline in Plasma Gamma-tocopherol (Vitamin E) at Day 7 From Day 0.
Description: Plasma measurements of gamma-tocopherol was assessed in response to smoking cessation and in combination with gamma-tocopherol (vitamin E) supplementation.
Time Frame: Day 0 and 7 of intervention
Measure: Mean (Standard Error); unit: microM
Arm/Group | Dietary Supplement + Smoking Cessation | Placebo + Smoking Cessation | Dietary Supplement + Nicotine Replacement Therapy | Placebo + Nicotine Replacement Therapy
Number analyzed (Participants) | 14 | 16 | 13 | 13
microM | 7.30 (0.98) | -0.10 (0.21) | 7.28 (1.57) | -0.24 (0.13)

3. Secondary Outcome: Absolute Change From Baseline in Plasma Malondialdehyde at Day 7 From Day 0.
Description: Plasma measurements of malondialdehyde, a marker of lipid peroxidation was assessed in response to smoking cessation and in combination with gamma-tocopherol (vitamin E) supplementation
Time Frame: Day 0 and 7 of intervention
Measure: Mean (Standard Error); unit: microM
Arm/Group | Dietary Supplement + Smoking Cessation | Placebo + Smoking Cessation | Dietary Supplement + Nicotine Replacement Therapy | Placebo + Nicotine Replacement Therapy
Number analyzed (Participants) | 14 | 16 | 13 | 13
microM | -0.08 (0.05) | -0.06 (0.03) | -0.04 (0.04) | -0.07 (0.02)

ADVERSE EVENTS:
Arm/Group | Dietary Supplement + Smoking Cessation | Placebo + Smoking Cessation | Dietary Supplement + Nicotine Replacement Therapy | Placebo + Nicotine Replacement Therapy
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/16 | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 0/14 | 0/16 | 0/13 | 0/13

LIMITATIONS AND CAVEATS:
Very few women were enrolled thereby precluding any assessment of potential gender differences for our outcome variables.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No